CLINICAL TRIAL: NCT07406269
Title: Evaluation of Clinical Effectiveness and Implementation of an Artificial Intelligence Based Decision Support Tool That Guides Early Rehabilitation After Gastrointestinal and Oncology Surgery
Brief Title: Clinical Evaluation of AI Decision Support for Early Rehabilitation After Surgery
Acronym: DESIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, D.E. Hilling, Surgeon and Data Scientist, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DESIRE implementation
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Oncologic Surgery; Gastrointestinal Cancers
Keywords: Artificial Intelligence; Clinical Decision Support System; Postoperative Care; Early Rehabilitation; Gastrointestinal Surgery; Oncological Surgery; Predictive Modeling
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cohort of 103 patients undergoing GE/oncological surgery and admitted >2 days after surgery (Experimental)
  Interventions: Device: DESIRE: AI-Based Clinical Decision Support for Postoperative Rehabilitation Planning

INTERVENTIONS:
Device: DESIRE: AI-Based Clinical Decision Support for Postoperative Rehabilitation Planning — The intervention consists of the clinical use of a locked, non-adaptive artificial intelligence (AI)-based clinical decision support system (DESIRE) that analyzes routinely collected electronic health record data to predict, on postoperative day 2, the risk that a patient will require hospital-specific interventions after gastrointestinal or oncological surgery.
  The system automatically extracts demographic, perioperative, vital sign, laboratory, and medication-related variables and generates a binary (yes/no) output indicating whether the patient is likely to be at low risk for requiring additional hospital care. A predefined conservative threshold is used to identify patients eligible for early rehabilitation.

SUMMARY:
After gastrointestinal or oncology surgery, it can be difficult to determine when a patient is ready to safely begin early rehabilitation or move toward discharge. Delays may prolong hospital stay, while premature decisions may increase risks.

This study evaluates an artificial intelligence (AI)-based decision support tool that analyzes routinely collected hospital data to identify patients who are likely ready for early rehabilitation and discharge planning after surgery. The tool provides a simple yes/no output to support clinicians in their decision-making.

The AI tool does not replace clinical judgment. Treating physicians remain fully responsible for all care decisions.

The purpose of this study is to examine how well this tool performs in clinical practice and how it can be safely and effectively implemented to support postoperative care.

DETAILED DESCRIPTION:
Patients who undergo gastrointestinal or oncology surgery often require careful monitoring after their operation. During the days following surgery, healthcare professionals assess many factors, such as vital signs, laboratory results, recovery progress, and the need for hospital-based treatments. Based on this information, decisions are made about when patients can safely start early rehabilitation or move toward discharge planning.

In this study, researchers are evaluating an artificial intelligence (AI)-based decision support tool designed to assist clinicians with these decisions. The tool analyzes routinely collected information from the electronic patient record, including demographic data, type of surgery, vital signs, laboratory values, and medication information. Using these data, the system provides a simple yes/no output indicating whether a patient is likely ready for early rehabilitation and discharge planning on the second day after surgery.

The AI tool is advisory only. It does not make treatment decisions and cannot initiate any actions. The treating physician always reviews the patient's condition independently and makes the final decision about care, rehabilitation, and discharge planning.

The study focuses on two main aspects:

1. How accurately the AI tool identifies patients who are ready for early rehabilitation and discharge planning.
2. How the tool can be safely and practically integrated into everyday clinical workflows.

Participation in this study does not change the standard of care. All patients continue to receive routine postoperative care according to existing hospital protocols. The AI tool serves solely as an additional source of information for clinicians.

Patient data used by the AI system are processed within secure hospital systems and handled in accordance with data protection regulations. No additional tests or procedures are required specifically for this study.

The results of this study may help improve postoperative care by supporting timely rehabilitation and discharge planning, potentially reducing unnecessary hospital stays while maintaining patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Undergoing gastrointestinal or oncological surgery
* Postoperatively admitted to the surgical ward
* Expected to remain admitted for at least 2 days after surgery

Exclusion Criteria:

* Admitted to the intensive care unit (ICU) at the time of prediction on postoperative day 2
* Inability to provide informed consent in Dutch or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients requiring unplanned escalation of hospital-specific care within 30 days after early transfer to rehabilitation area. | From postoperative day 2 (time of AI prediction and potential transfer to rehabilitation area) through 30 days after surgery
  This is a composite outcome, consisting of any of the following events:
  ICU admission
  Re-operation
  Radiological intervention
  Administration of intravenous antibiotics
  Respiratory failure (new need for supplemental oxygen)
  30-day mortality
  30-day emergency readmission

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided